CLINICAL TRIAL: NCT04696692
Title: Single-Cell Map of Immune and Lymphoma Cells in B-cell Non-Hodgkin's Lymphoma
Acronym: SIMILY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20 HEMA 10
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: Diffuse large B-cell lymphoma; R-CHOP treatment; Biomarker; Single-cell sequencing
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with histologically confirmed diffuse large B-cell lymphoma (Other)
  Interventions: Other: Patient with histologically confirmed diffuse large B-cell lymphoma with a planned first line treatment by R-CHOP.

INTERVENTIONS:
Other: Patient with histologically confirmed diffuse large B-cell lymphoma with a planned first line treatment by R-CHOP. — Blood samples will be collected :
  * at baseline (before the 1st R-CHOP cycle)
  * before the 3d administration of chemotherapy (CT) (i.e. after 2 cycles of CT and same timepoint as interim FDG-PET/CT)
  * after the 4th administration of the CT
  * at the end of induction (i.e. end of R-CHOP treatment)
  * at 24 months after initiation of R-CHOP treatment
  * at the time of progression (if progression occurs before 24 months of treatment).
  Tumor samples will be collected at baseline (from an archived initial diagnostic tumor specimen) and at the time of progression (if applicable from lymph node biopsy performed as part of a standard of care surgical procedure).
  Bone marrow samples will be collected at baseline and at the time of progression (if applicable) only in patients for whom a bone marrow aspiration (BMA) is necessary as part of their standard of care, upon physician's decision.

SUMMARY:
This trial is a translational, prospective, open-label, monocentric research.

The study will be conducted in a population of 60 patients with diffuse large B-cell lymphoma (DLBCL) for whom first-line treatment with R-CHOP is planned as part of their standard of care.

SIMILY program aims at identifying biomarkers and/or molecular signatures related to immuno-phenotypic and -genotypic characteristics of the tumor and immune microenvironment, at the time of diagnosis, during R-CHOP, and at 24 months or time of progression.

Each patient will be followed during 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with histologically confirmed diffuse large B-cell lymphoma with a planned first line treatment by R-CHOP (treatment by R-CHOP should not have been initiated prior to inclusion in the study)
2. Age 18 to 80 years at the time of study entry
3. Archived initial diagnostic tumor specimen available
4. Life expectancy ≥ 3months
5. ECOG Performance status 0-2
6. FDG-avid disease (for PET monitoring)
7. Signed written informed consent
8. Patient able to participate and willing to give informed consent prior performance of any study-related procedures and to comply with the study protocol
9. Patient affiliated to a Social Health Insurance in France

Exclusion Criteria:

1. Patient pregnant, or breast-feeding
2. Any condition contraindicated with tumor / blood sampling procedures required by the protocol
3. Central Nervous System (CNS) involvement
4. Known history of positive test for Hepatitis B virus or Hepatitis C virus or Immunodeficiency Virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
5. Any current severe or uncontrolled disease, including, but not limited to ongoing or active infection and auto immune disorders
6. Any psychological, familial, geographic or social situation, according to the judgment of investigator, potentially preventing the provision of informed consent or compliance to study procedure
7. Patient who has forfeited his/her freedom by administrative or legal award or who is under legal protection (curatorship and guardianship, protection of justice)
8. Current participation in any other therapeutic clinical study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2025-12-11 (Actual); Study Completion 2025-12-11 (Actual)

PRIMARY OUTCOMES:
Levels of ctDNA to determine if it reflect the disease evolution of patient with DLBCL treated in first line. | 24 months for each patient
Levels of tumor tissue biomarkers to determine if it reflect the disease evolution of patient with DLBCL treated in first line. | 24 months for each patient
  Tumor tissue biomarkers will be identified by ScRNA sequencing and targeted NGS.
Levels of blood biomarkers to determine if it reflect the disease evolution of patient with DLBCL treated in first line. | 24 months for each patient
  Blood biomarkers will be identified by ScRNA sequencing.

SECONDARY OUTCOMES:
Levels of tumor tissue biomarkers compared to clinical data in the prediction of treatment response. | 24 months for each patient
  Tumor tissue biomarkers will be identified by ScRNA sequencing and targeted NGS.
Levels of blood biomarkers compared to clinical data in the prediction of treatment response. | 24 months for each patient
  Blood biomarkers will be identified by ScRNA sequencing.
Levels of ctDNA compared to conventional PET imaging (at the standard time points) in the prediction of treatment response. | 24 months for each patient

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Universitaire du Cancer Toulouse - Oncopole, Toulouse, France